CLINICAL TRIAL: NCT00082329
Title: Peripheral Blood Hematopoietic Progenitor Cell Mobilization Using Granulocyte Colony Stimulating Factor (G-CSF) Combined With AMD3100 Mozobil (Plerixafor) in Healthy Volunteers
Brief Title: G-CSF and AMD3100 to Mobilize Stem Cells in Healthy Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040179; 04-H-0179 (Other: NIH NHLBI)
Record Dates: First submitted 2004-05-06; First posted 2004-05-06 (Estimated); Results first posted 2014-05-02 (Estimated); Last update posted 2021-07-22 (Actual); Status verified 2021-05

CONDITIONS: Healthy
Keywords: Hematopoietic Stem Cells; PBSC's; Mobilization; Alloreactivity; T Cell Polarization; Dendritic Cells; CXCR4; Plerixafor; Healthy Volunteer (HV)
MeSH Terms: interventions — plerixafor; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- G-CSF and AMD3100 to Mobilize Stem Cells in Healthy Volunteers (Experimental): Participants received subcutaneous injection of G-CSF (10 mcg/kg/day) for 5 days followed by a single subcutaneous injection of AMD3100 (240 mcg/kg) given 12 hours prior to apheresis peripheral blood stem cell collection. Peripheral blood stem cell collection performed on the fifth day of G-CSF administration.
  Interventions: Drug: AMD 3100 (Mozobil plerixafor); Drug: Granulocyte colony-stimulating factor (G-CSF)

INTERVENTIONS:
Drug: AMD 3100 (Mozobil plerixafor) — Participants received subcutaneous injection of granulocyte colony-stimulating factor (G-CSF) at 10 mcg/kg/day for 5 days followed by a single subcutaneous injection of AMD3100 (240 mcg/kg) given 12 hours prior to apheresis peripheral blood stem cell collection. Peripheral blood stem cell collection performed on the fifth day of G-CSF administration.
  Other Names: AMD 3100
Drug: Granulocyte colony-stimulating factor (G-CSF) — Participants received subcutaneous injection of granulocyte colony-stimulating factor (G-CSF) at 10 mcg/kg/day for 5 days followed by a single subcutaneous injection of AMD3100 (240 mcg/kg) given 12 hours prior to apheresis peripheral blood stem cell collection. Peripheral blood stem cell collection performed on the fifth day of G-CSF administration.
  Other Names: G-CSF

SUMMARY:
This 12-day study will test whether the combination of G-CSF (granulocyte-colony stimulating factor) and AMD3100 (Mozobil) is more efficient in mobilizing stem cells for collection than the use of G-CSF alone. Traditionally, the growth factor G-CSF has been given to stem cell donors to mobilize, or push, stem cells out of the bone marrow and into the blood circulation for collection for transplantation. Although a sufficient quantity of cells usually can be collected with G-CSF treatment, some donors do not respond well and may require multiple apheresis procedures (see below) to collect enough cells. Studies indicate that G-CSF used together with a drug called AMD3100 may be more effective in mobilizing stem cells for collection than G-CSF alone. The Food and Drug Administration has approved G-CSF for stem cell mobilization. AMD3100 is a new drug that also mobilizes stem cells in large numbers within a few hours.

Normal healthy volunteers between 18 and 60 years of age may be eligible for this study.

DETAILED DESCRIPTION:
Peripheral blood progenitor cells (PBPC) are the most popular source of hematopoetic stem cells for allogeneic transplantation because of technical ease of collection and faster engraftment. Traditionally, granulocyte-colony stimulating factor (G-CSF) has been used to procure the peripheral blood stem cell graft. Although regimens using G-CSF usually succeed in collecting adequate numbers of PBPC from healthy donors, 5%-10% of the donors will mobilize stem cells poorly and may require multiple large volume apheresis or bone marrow harvesting. AMD3100 reversibly inhibits CXC- chemokine receptor 4 (CXCR4) binding to stromal cell derived factor (SDF) - 1 and was recently discovered to be an effective agent to mobilize cluster of differentiation 34 (CD34)+ cells into the peripheral blood. In normal volunteers, administering AMD3100 after 4-5 days of G-CSF resulted in a 3-3.5 fold increase in circulating CD34 cells compared to G-CSF alone. Recent data has suggested that the combination of G-CSF and AMD3100 is superior to G-CSF alone for mobilizing hematopoietic progenitor cells in heavily pretreated patients with multiple myeloma or non-Hodgkin's lymphoma undergoing autologous hematopoietic transplantation. Combining AMD3100 with G-CSF could be an effective strategy to improve the yield of PBPC collected from allogeneic donors who mobilize poorly with G-CSF alone. However, the biological impact of AMD3100 in this context on T cells and other cellular populations contained within the allograft that mediate graft versus host disease (GVHD) and graft-versus-leukemia (GVL) effects are unknown.

We propose to collect peripheral progenitor cell (PBPC) from healthy volunteers following 5 days of G-CSF (10 mcg/kg/day) and a single dose of AMD3100 (240 mcg/kg subcutaneous given 12 hours before starting apheresis) to study the impact of combining these two mobilizing agents on the immunological properties of the mobilized cells. A single 15 liter apheresis will be conducted on day 5 following the 5th dose of G-CSF. The immunological studies conducted on these mobilized cells will be the same as our parallel study which is investigating the immune properties of PBPCs mobilized with G-CSF or AMD3100 alone. If combining AMD3100 with G-CSF has no negative impact on the immune populations involved in GVHD and graft-vs-leukemia effects, this regimen could be used for allogeneic donors who fail to mobilize sufficient peripheral blood stem cell (PBSC) using G-CSF alone.

Primary objective: To determine the cytokine polarization status of cluster of differentiation 4 (CD4+) T-cells collected by apheresis following combination of AMD3100 and G-CSF compared to G-CSF mobilization.

Primary endpoint: the ratio of Th1 [intracellular interferon (IFN-g) +] versus Th2 [intracellular interleukin (IL-4+)] T-cells in the apheresis products collected from individual donors undergoing mobilization with combination of G-CSF and AMD3100 to the ratio in apheresis product collected with G-CSF alone (ratio published in literature).

Secondary endpoints: To examine 1) the cellular content and other immune properties of mobilized cells; 2) yields of hematopoietic progenitor cells, immune cells, and other cellular subsets collected by apheresis; and the 3) safety profile of AMD3100.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy volunteers greater or equal to 18 years old, less than or equal to 60 years.

Weight greater than 60 kg (132 pounds)

Normal renal function: creatinine less than 1.5 mg/dl l

Normal liver function: bilirubin less than1.5mg/dl, transaminases within normal limit

Normal blood count: white blood cell (WBC) 3000-10000/mm3, granulocytes greater than 1500/mm3, platelets greater than 150,000/mm3, hemoglobin greater than 12.5g/dl

Subject must be eligible for normal blood donation and fit to undergo apheresis procedure (antecubital veins must be adequate for peripheral access during apheresis)

Ability to comprehend the investigational nature of the study and provide informed consent

EXCLUSION CRITERIA: any of the following

Active infection or history of recurrent infection or positive test for syphilis (RPR), hepatitis B and C (HBaSAg, Anti-HCV), HIV and human T- Lymphocytic virus (HTLV-1)

History of autoimmune disease such as rheumatoid arthritis, systemic lupus erythematous

History of cancer within the past 5 years excluding basal cell or squamous cell carcinoma of the skin

History of any hematologic disorders including thromboembolic disease

History of cardiac disease such as uncontrolled hypertension, peripheral vascular disease, myocardial infarction, cardiac arrhythmias or related symptoms such as tachycardia, chest pain, shortness of breath which have required medical intervention or treatment or a Framingham coronary disease risk prediction score of greater than 10% 10 year coronary heart disease (CHD) risk

History of heavy smoking with underlying pulmonary disease

History of cerebrovascular disease, transient ischemic attack, or stroke

Diagnosis of sickle cell anemia or sickle cell trait (to be screened by hemoglobin (Hbg) electrophoresis)

Pregnant or lactating

Severe psychiatric illness: mental deficiency sufficiently severe as to make informed consent impossible.

Mobilization with G-CSF within 90 days of protocol enrollment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2004-06-18 (Actual); Primary Completion 2012-10-25 (Actual); Study Completion 2012-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Childs, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gyger M, Stuart RK, Perreault C. Immunobiology of allogeneic peripheral blood mononuclear cells mobilized with granulocyte-colony stimulating factor. Bone Marrow Transplant. 2000 Jul;26(1):1-16. doi: 10.1038/sj.bmt.1702464. PMID 10918400
- [Background] Bellucci R, De Propris MS, Buccisano F, Lisci A, Leone G, Tabilio A, de Fabritiis P. Modulation of VLA-4 and L-selectin expression on normal CD34+ cells during mobilization with G-CSF. Bone Marrow Transplant. 1999 Jan;23(1):1-8. doi: 10.1038/sj.bmt.1701522. PMID 10037043
- [Background] Mohle R, Murea S, Kirsch M, Haas R. Differential expression of L-selectin, VLA-4, and LFA-1 on CD34+ progenitor cells from bone marrow and peripheral blood during G-CSF-enhanced recovery. Exp Hematol. 1995 Dec;23(14):1535-42. PMID 8542944
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2004-H-0179.html

RESULTS

PARTICIPANT FLOW:
Groups:
- G-CSF and AMD3100 to Mobilize Stem Cells in Healthy Volunteers: Participants received subcutaneous injection of granulocyte colony-stimulating factor (G-CSF) at 10 mcg/kg/day for 5 days followed by a single subcutaneous injection of AMD3100 (240 mcg/kg) given 12 hours prior to apheresis peripheral blood stem cell collection. Peripheral blood stem cell collection was performed on the fifth day following G-CSF administration.
Period: Overall Study
Arm/Group | G-CSF and AMD3100 to Mobilize Stem Cells in Healthy Volunteers
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | G-CSF and AMD3100 to Mobilize Stem Cells in Healthy Volunteers
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Apheresis Collection Following Combination of AMD3100 and G-CSF.
Description: Healthy volunteers will be administered AMD 3100 (Mozobil plerixafor) and granulocyte colony stimulating factor (G-CSF) to determine cytokine polarization status of cluster of differentiation (CD 4) T-cells collected by apheresis.
  We propose that the combination of single dose AMD 3100 and G-CSF as combined mobilizing agents will improve the peripheral blood progenitor cells mobilization. Successful treatment responders is defined by completing study treatment with cell mobilization and cell collection. Non-responders is defined by having completed the study treatment and having cell mobilization without cell collection.
Time Frame: Day 1 (cells are counted 24 hours after AMD3100)
Measure: Number; unit: participants
Arm/Group | G-CSF and AMD3100 to Mobilize Stem Cells in Healthy Volunteers
Number analyzed (Participants) | 9
participants
  AMD & G-CSF Responder | 8
  AMD& G-CSF Non-Responder | 1

2. Secondary Outcome: Average Fold Change From Baseline of Mobilized Cells Following G-CSF and AMD3100 to Mobilize Stem Cells in Healthy Volunteers
Description: Average fold change from baseline of mobilized cells that contained immune properties and other cellular content following G-CSF and AMD3100 to mobilize stem cells in healthy volunteers. The mobilized cells are defined as: white blood cells, lymphocytes, polys and monocytes. Polys (also known as segs, segmented neutrophils, neutrophils, granulocytes) are the most numerous of our white blood cells.
Time Frame: Day 7
Measure: Mean (Full Range); unit: Mean Fold Change from Baseline
Arm/Group | G-CSF and AMD3100 to Mobilize Stem Cells in Healthy Volunteers
Number analyzed (Participants) | 9
Mean Fold Change from Baseline
  White Blood Cells | 9.3 [6.6 to 14]
  Lymphocytes | 3.8 [2.4 to 5.3]
  Polys | 11.9 [7.2 to 17.8]
  Monocytes | 6.6 [2.2 to 12.2]

3. Secondary Outcome: Number of Participants With Increased the Levels of Circulating Hematopoietic Progenitor Cells, Immune Cells, and Other Cellular Subsets Collected by Apheresis.
Description: Number of participants with increase in yields of hematopoietic progenitor cells, immune cells, and other cellular subsets collected by apheresis following G-CSF and AMD3100 to mobilize stem cells.
Time Frame: Day 7
Population: 1 participant did not complete apheresis, therefore 1 participant was not included in analysis
Measure: Number; unit: participants
Arm/Group | G-CSF and AMD3100 to Mobilize Stem Cells in Healthy Volunteers
Number analyzed (Participants) | 9
participants | 8

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | G-CSF and AMD3100 to Mobilize Stem Cells in Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | G-CSF and AMD3100 to Mobilize Stem Cells in Healthy Volunteers (N=9)
deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | G-CSF and AMD3100 to Mobilize Stem Cells in Healthy Volunteers (N=9)
Elevated Alk Phos (Blood and lymphatic system disorders) | 8
Elevated LDH (Blood and lymphatic system disorders) | 8
Elevated WBCs (Blood and lymphatic system disorders) | 1
tachycardia (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
achy (General disorders) | 1
Appetite decr'd (General disorders) | 1
Body ache (General disorders) | 1
diaphoresis (General disorders) | 1
fatigue (General disorders) | 3
Headache (General disorders) | 3
low back pain (General disorders) | 1
Tiredness (General disorders) | 1
Tiredness (fatigue) (General disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1
bone pain (Musculoskeletal and connective tissue disorders) | 3
low back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle pain (Musculoskeletal and connective tissue disorders) | 1
paresthia (facial tingling) (Nervous system disorders) | 1
Mood alteration (Psychiatric disorders) | 1
Bruising, local at IV site (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No